CLINICAL TRIAL: NCT02223247
Title: A Phase 1, First-In-Human Study of Escalating Doses of Oral TVB-2640 in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sagimet Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3V2640-CLIN-002
Record Dates: First submitted 2014-08-18; First posted 2014-08-22 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Solid Malignant Tumor
Keywords: solid tumors; cancer
MeSH Terms: conditions — Neoplasms | interventions — TVB-2640

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TVB-2640 (Experimental): Oral TVB-2640 capsules or tablets of various dose strengths administered QD for 21 - 28 day dosing cycles, alone or in combination with certain standard chemotherapy agents
  Interventions: Drug: TVB-2640

INTERVENTIONS:
Drug: TVB-2640

SUMMARY:
This first in human phase 1 study of TVB-2640 is being conducted in patients with advanced stage solid malignant tumors. This research is being done to find out how safe and useful TVB-2640 is for patients who have received previous cancer therapy, and for whom no therapy exists that would be curative or might provide significant benefit. TVB-2640 belongs to a class of drugs called fatty acid synthase inhibitors (FASN inhibitors). This means that they interfere with the body's (and the tumor's) ability to use a substance called fatty acid synthase (FASN). Research has shown that some tumors appear to need FASN to keep growing.

ELIGIBILITY:
Inclusion Criteria Include:

* Patient has histologically- or cytologically- confirmed metastatic or advanced-stage solid malignant tumor that is refractory to standard therapy and for whom no therapy exists that would be curative or might provide significant benefit and therefore for whom experimental therapy is a reasonable option.
* Patient experienced progressive disease during or following or was intolerant of their most recent treatment regimen.
* Patient is male or female aged ≥18 years.
* Patient has an ECOG performance status of 0 (fully active, able to carry out all pre-disease activities without restriction) or 1 (unable to perform physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature), as assessed on C1D1, before the first dose of TVB 2640.
* Patient has adequate renal function (creatinine ≤1.5 times the upper limit of normal [ULN]) or a glomerular filtration rate (GFR) of ≥50 mL/min.
* Patient has adequate hepatic function,
* Patient has adequate bone marrow function
* Patient has no significant ischemic heart disease or myocardial infarction (MI) within 6 months before the first dose of TVB 2640 and currently has adequate cardiac function

For the Monotherapy Expansion Cohorts of the Study ONLY:

* Patient has a specific tumor-type and histology, as designated by the Sponsor based on nonclinical and clinical data obtained prior to enrollment in the Expansion Cohort.
* Patient has measurable disease, as determined by the Investigator using RECIST, version 1.1 (1).

For the Combination Cohorts ONLY:

* In addition to meeting monotherapy criteria above, the commercially-available anticancer agent of interest being investigated in combination with TVB-2640, administered according to the dose regimen in the prescribing information, is deemed appropriate for the patient's disease and clinical status.

Exclusion Criteria Include:

* Patient is unable to swallow oral medications or has impairment of GI function or GI disease that may significantly alter drug absorption
* Patient has uncontrolled or severe intercurrent medical condition (including uncontrolled brain metastases).
* Patient underwent major surgery within 4 weeks before the first dose of TVB 2640 or received cancer-directed therapy or an investigational drug or device within 4 weeks (6 weeks for mitomycin C and nitrosoureas) or 5 half-lives of that agent (whichever is shorter) before the first dose of TVB 2640.
* If female, patient is pregnant or breast-feeding.
* Patient has evidence of a serious active infection
* Patient has a history of other malignancy treated with curative intent within the previous 5 years with the exception of adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) based on toxicity analysis. | 1.5 years
  Toxicity will be monitored according to NCI - Common Toxicity Criteria for Adverse Events version (4.03). Patients receiving at least one dose of drug.
To determine the incidence and nature of dose-limiting toxicities (DLTs) of TVB-2640. | Days 1 to 21 of cycle 1 for monotherapy cohort(s); Days 1 to 28 of cycle 1 for combination with anti-cancer agent cohort(s)

SECONDARY OUTCOMES:
Incidence, nature and severity of adverse events and serious adverse events, graded according to NCI - Common Toxicity Criteria for Adverse Events version (4.03). | Up to 28 days after the last dose of study treatment or until initiation of another anti-cancer therapy, whichever occurs first.
Pharmacokinetic parameters of TVB-2640 (including total exposure, maximum and minimum serum concentration, clearance, volume of distribution at steady state) | At Cycle Day 1, 2, 8, 15, (and 22 for combination cohorts) then the first day of subsequent cycles until discontinuation.
  Cmax, Cmin, Tmax, AUC and Half-life of TVB-2640
Tumor response per RECIST 1.1 | Measured every 6 weeks for 21 day cycles or every 8 weeks for 28 day cycles for the duration of study treatment, estimated to be less than one year

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Infante, MD, Principal Investigator — The Sarah Cannon Research Institute
Locations (11):
- United States (7):
  - Scottsdale, Arizona
  - Denver, Colorado
  - Sarasota, Florida
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
- United Kingdom (4):
  - Charthouse Square, London
  - London
  - Manchester
  - West Smithfield, London

REFERENCES:
- [Derived] Falchook G, Infante J, Arkenau HT, Patel MR, Dean E, Borazanci E, Brenner A, Cook N, Lopez J, Pant S, Frankel A, Schmid P, Moore K, McCulloch W, Grimmer K, O'Farrell M, Kemble G, Burris H. First-in-human study of the safety, pharmacokinetics, and pharmacodynamics of first-in-class fatty acid synthase inhibitor TVB-2640 alone and with a taxane in advanced tumors. EClinicalMedicine. 2021 Mar 30;34:100797. doi: 10.1016/j.eclinm.2021.100797. eCollection 2021 Apr. PMID 33870151